CLINICAL TRIAL: NCT02581696
Title: An Open-label, Multiple-dose, Single-arm, Phase 1 Study to Evaluate the Drug-drug Interaction and Safety of Lafutidine and Irsogladine Maleate in Healthy Adult Volunteers
Brief Title: The Drug-drug Interaction and Safety of Lafutidine and Irsogladine Maleate in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BR-LAF-CT-101
Record Dates: First submitted 2015-10-12; First posted 2015-10-21 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Peptic Ulcer
MeSH Terms: conditions — Peptic Ulcer | interventions — lafutidine; irsogladine

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): This is a follow-up study of BR-LAF-CT-101, a phase 1 study to evaluate the drug-drug interaction and safety of Lafutidine and Irsogladine maleate in healthy adult volunteers. Subjects judged to be appropriate to this study by screening.
  Interventions: Drug: Lafutidine; Drug: Irsogladine maleate

INTERVENTIONS:
Drug: Lafutidine — Lafutidine 10mg, 1 tablet, bid
  Other Names: STOGAR
Drug: Irsogladine maleate — Irsogladine maleate 2mg, 2 tablet, qd
  Other Names: STOWON

SUMMARY:
An open-label, multiple-dose, single-arm, phase 1 study to evaluate the drug-drug interaction and safety of Lafutidine and Irsogladine maleate in healthy adult volunteers

DETAILED DESCRIPTION:
A phase 1 study to evaluate the drug-drug interaction and safety of Lafutidine and Irsogladine maleate in healthy adult volunteers. Subjects judged to be appropriate to this study by screening before 28days of first administration. Subjects administrate Lafutidine bid during period I. After wash-out period, administrate Irsogladine maleate qd during Period II. After than, coadministration Lafutidine bid and Irsogladine maleate qd.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between the ages of 19 and 50 at the screening
2. Male subjects whose weight is greater than 55kg Female subjects whose weight is greater than 50kg and within ±20% range of ideal body weight.

   Ideal body weight(kg) = (Height(cm) - 100) * 0.9
3. For female subjects must show negative for urine pregnancy test and also must meet one of the below listed criteria:

   * A menopausal woman (Menstruation should stop at least 2 years ago)
   * Take sterilization operation (Hysterectomy, Ovariotomy, Tubal ligation, any other operation)
   * Male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for the female subject.
   * Before 3 months of the screening and 1month after the end of drug administration, subjects must meet contraception requirements.
   * For avoiding the drug-drug interaction, subjects must not use any contraceptive drugs and must choose abstinence or use physical block.
4. A sexually active male subjects must use and accepted method of contraception during the course of the clinical study and must not donate sperms until a month after finishing drug administration. (If male subjects oneself or female partner is sterility, that does not apply.)
5. Subjects who understand the clinical study completely, agree to participate and sign written consent form for conduct precautions

Exclusion Criteria:

1. Subjects having liver system disorders, kidney disorders, digestive system disorders, cardiovascular disorders, respiratory disorders, endocrine disorders, neurological disorder or hematological disorders, psychiatric disorders, or a history of malignancy, disorders
2. Subjects having a history of gastrointestinal system disorders influencing drug absorption(i.e, Crohn's disease, ulcer) or surgery (except simple typhlectomy or hernia repair surgery)
3. Subjects having a history of hypersensitivity to additional ingredient or clinically significant hypersensitivity to lafutidine and Irsogladine or any other drug.
4. Subjects who judged for inappropriate to physical examination. ( Disease history, physical examine, vital sign, EKG examine, laboratory examine and so on ).
5. Galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption and any other hereditary disorder.
6. Subjects who is sitting after 5minutes break, having Systolic blood pressure ≥ 140 mmHg and Diastolic blood pressure ≤ 90 mmHg, or Systolic blood pressure ≥ 90 mmHg and Diastolic blood pressure ≤ 60 mmHg on vital sign
7. Subjects having a history of drug abuse or positive drug abuse urinalysis testing at screening.
8. Subjects who is pregnancy or feed breast milk.
9. Subjects who has participated in another clinical study before study drug administration Subjects having blood donation within two months or component blood donation within one month before study drug administration
10. Subjects who has drunken beverages caffeine-containing or alcohol or smoking during prohibition period
11. Subjects who has judged to be inappropriate for this study by investigators according to other reasons including clinical lab test result

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve of Lafutidine and Irsogladine maleate | Sampling time 1, 19, 21days before drug administration, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hr after drug administration. (total 24times)

SECONDARY OUTCOMES:
Peak Plasma Concentration of Lafutidine and Irsogladine | Sampling time 1, 19, 21days before drug administration, and 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24hr after drug administration. (total 24times)

CONTACTS AND LOCATIONS:
Overall Officials: Seoung-hun Han, Professor, Principal Investigator — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No